CLINICAL TRIAL: NCT00006073
Title: Endocrine Studies in Health and Disease
Status: Terminated | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000180; 00-CH-0180
Record Dates: First submitted 2000-07-25; First posted 2003-07-14 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-08-31

CONDITIONS: Endocrine Diseases
Keywords: Evaluation; Endocrinology; Hormones; Metabolism; Teaching; Endocrine Disorder
MeSH Terms: conditions — Endocrine System Diseases

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will evaluate healthy normal volunteers and patients with a variety of endocrine disorders to 1) learn more about conditions that affect the endocrine glands (glands that secrete hormones) and 2) train physicians in endocrinology.

Patients with endocrine-related conditions and healthy volunteers of all ages may be eligible for this study.

All participants will have a physical examination medical and history. They may be required to provide blood, saliva or urine samples and undergo ultrasound (using sound waves) or magnetic resonance (using a magnetic field) imaging to visualize internal body structures.

Some healthy adult volunteers will have hormone-stimulating tests to assess endocrine function. These tests measure blood hormone levels before and after injection of a synthetic form of a hormone. A device called a heparin lock, through which the hormone is injected and the blood samples are collected, is placed in a vein in the arm or hand. Blood samples are drawn before the hormone is injected and at various intervals after the injection to measure levels of the hormone. These tests, which last from 1 to 3 hours, may include the following:

1. CRH stimulation test corticotropin-releasing hormone is given to test pituitary and adrenal gland function
2. ACTH stimulation test adrenocorticotrophic hormone is given to test adrenal gland function
3. LHRH stimulation test luteinizing hormone-releasing hormone is given to test pituitary gland function
4. TRH stimulation test thyroid-releasing hormone is given to test pituitary and thyroid gland function
5. GHRH stimulation test growth hormone releasing hormone is given to measure growth hormone levels.

An oral glucose tolerance test, which is similar to the stimulation tests, may also be done to measure blood glucose (sugar) and insulin levels after drinking a sugary liquid.

Healthy volunteers and patients with a hereditary endocrine disorder and their family members may also be asked to provide a blood sample for genetic studies of inherited endocrine disorders. Patients with endocrine-related disorders may be offered medical or surgical treatment for their disorder.

AcAccess http://turners.nichd.nih.gov/ for additional study publications.

DETAILED DESCRIPTION:
This protocol is designed to allow endocrine-related evaluations of healthy subjects and patients with a variety of endocrine disorders. Healthy subjects may be studied to obtain normative data for endocrine tests involving blood, urine, saliva, ultrasound and magnetic resonance examinations. If not eligible for a specific NICHD research protocol, patients with endocrine-related conditions may be evaluated under the auspices of this protocol to advance the clinical skills of physicians participating in NICHD clinical research and training programs, and to provide stimuli for new clinical research initiatives. Standard, medically-indicated laboratory or radiological studies may be performed to confirm a diagnosis or to aid in the management of the patient. In some cases, the patient will receive medical or surgical treatment for their disorder, according to current clinical practice. The overall purpose of endocrine evaluations under this protocol is to support our clinical training and research missions.

ELIGIBILITY:
* INCLUSION CRITERIA

Healthy subjects and patients with endocrine-related conditions of all ages are eligible for this protocol. The actual selection of patients most appropriate for clinical training needs will be made by protocol investigators.

Subjects with disabilities are not formally excluded from the study unless the disability would specifically prevent their participation. If a subject with cognitive impairment wishes to participate, there must be available a family member or other qualified individual holding a durable power of attorney who is able to guide the impaired subject s participation and be an advocate for their interests. This participation is limited to the non-research, clinical training arm of the study.

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3090 (Actual)
Dates: Start 2000-07-19; Study Completion 2016-08-31

CONTACTS AND LOCATIONS:
Overall Officials: Margaret F Keil, C.R.N.P., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Han JC, Reyes-Capo DP, Liu CY, Reynolds JC, Turkbey E, Turkbey IB, Bryant J, Marshall JD, Naggert JK, Gahl WA, Yanovski JA, Gunay-Aygun M. Comprehensive Endocrine-Metabolic Evaluation of Patients With Alstrom Syndrome Compared With BMI-Matched Controls. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2707-2719. doi: 10.1210/jc.2018-00496. PMID 29718281